CLINICAL TRIAL: NCT00408759
Title: Phase 2 Study of Hypnosis for Treating Xerostomia Following Radiotherapy in Head & Neck Cancer Patients
Brief Title: Hypnosis for Treating Xerostomia Following Radiotherapy in Head & Neck Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eschiff
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2006-12-07 (Estimated); Status verified 2006-12

CONDITIONS: Xerostomia
Keywords: xerostomia; hypnosis; dry mouth; radiotherapy; head and neck cancer
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms | interventions — Hypnosis

INTERVENTIONS:
Behavioral: hypnosis

SUMMARY:
xerostomia develops in all patients with head and neck cancer following radiotherapy. it consists one of the main side effects which affects quality of life. currently, there is no standard of care for treating this condition. parasympathomimetic drugs may help but carry significant side effects.

hypnosis may affect autonomic function such as salivation, in healthy people.in this study we will explore the efficacy of hypnosis in improving salivation, in the patient population.

DETAILED DESCRIPTION:
10 head and neck cancer patients with xerostomia following radiotherapy will be assessed for severity of xerostomia using questionnares and quantitative salivation tests. patients responsive to citric acid will receive a hypnotic session with specific suggestion for salivation. saliva volume will be assessed pre and post hypnosis. patients will receive a CD with recorded hypnotic session to use freely at home. xerostomia will be assessed using a questionnare one week following hypnosis.

ELIGIBILITY:
Inclusion Criteria:

* radiotherapy for head and neck cancer
* xerostomia

Exclusion Criteria:

* psychiatric illness (present or past)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-11; Study Completion 2006-12

PRIMARY OUTCOMES:
salivaa volume
quality of life related to salivation

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, Principal Investigator — Bnai Zion MC
Locations (1):
- bnai zion MC, Haifa, Israel